CLINICAL TRIAL: NCT01505374
Title: Saphenous Nerve Block vs. Femoral Nerve Block for Total Knee Arthroplasty: A Comparative Effectiveness Study in Bilateral Total Knee Arthroplasty Patients
Brief Title: Saphenous Nerve Block vs. Femoral Nerve Block for Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2012-033
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Difference Between Femoral Nerve Block and Saphenous Block
Keywords: Bilateral total knee replacement; Femoral Nerve Block; Saphenous Nerve Block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Technique Left Leg, Control Technique Right Leg (Experimental)
  Interventions: Procedure: Study Technique; Procedure: Control Technique
- Study Technique Right Leg, Control Technique Left Leg (Experimental)
  Interventions: Procedure: Study Technique; Procedure: Control Technique

INTERVENTIONS:
Procedure: Study Technique — One leg will receive the saphenous nerve block, at the level of the adductor canal (study technique). The block will be under ultrasound guidance. The local anesthetic will be 15 ml of 0.5% bupivacaine. All study patients, regardless of study arm will receive combined spinal epidural, with 3 ml of 0.5% bupivacaine as the spinal agent. Epidural local anesthetic, if needed, will consist of 2% lidocaine.
Procedure: Control Technique — The other leg will receive the femoral nerve block (control technique). The block will be under ultrasound guidance. The local anesthetic will be 30 ml of 0.25% bupivacaine. All study patients, regardless of study arm will receive combined spinal epidural, with 3 ml of 0.5% bupivacaine as the spinal agent. Epidural local anesthetic, if needed, will consist of 2% lidocaine.

SUMMARY:
Currently, the regional anesthetic standard of care for total knee replacement surgery is combined spinal/epidural to provide long-lasting pain relief with or without a femoral nerve block (FNB). The femoral nerve block refers to a technique that your anesthesiologist can use to numb the thigh muscle for approximately 18 hours after surgery. While this technique offers significant pain relief, it is possible it may cause muscle weakness and increase patients' recovery times. Hence there is a need for an alterative anesthetic technique, one that may help minimize postoperative pain as effectively as a femoral nerve block, while not causing weakness of the thigh muscle.

The saphenous nerve, a branch of the femoral nerve, provides sensation to the knee. Thus it is hypothesized by "blocking" or anesthetizing the saphenous nerve with local anesthetic closer to where it branches off, the area around and below the knee will feel numb. Yet unlike the femoral nerve block, the thigh muscle itself will still be able to function.

For patients undergoing two total knee replacements at one time or bilateral total knee replacement, they will be randomly assigned to receive a femoral nerve block on one leg and a saphenous block on the other. Pain levels will be measured and thigh muscle strength will be tested using a dynamometer before surgery, 6-8 hours following anesthesia administration, and on postoperative days 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* All patients ages 40-80 undergoing Bilateral Total Knee Replacement
* Planned use of neuraxial anesthesia
* Ability to follow study protocol

Exclusion Criteria:

* Contraindication to a spinal or epidural anesthestic
* Not a candidate for bilateral total knee replacement
* Chronic opioid use (defined as daily or almost daily use of opioids for >3 months)
* Hypersensitivity and/or allergy to local anesthetics
* Intraoperative use of any volatile anesthetic
* Patients with pre-existing neuropathy on the operative limb
* Contraindication to femoral nerve block or saphenous nerve block
* Allergy to any of the study medications
* American Society of Anesthesiologists (ASA) Class 4-5
* Non-English speaking patients

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stavros G. Memtsoudis, MD, PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Capdevila X, Barthelet Y, Biboulet P, Ryckwaert Y, Rubenovitch J, d'Athis F. Effects of perioperative analgesic technique on the surgical outcome and duration of rehabilitation after major knee surgery. Anesthesiology. 1999 Jul;91(1):8-15. doi: 10.1097/00000542-199907000-00006. PMID 10422923
- [Background] Singelyn FJ, Ferrant T, Malisse MF, Joris D. Effects of intravenous patient-controlled analgesia with morphine, continuous epidural analgesia, and continuous femoral nerve sheath block on rehabilitation after unilateral total-hip arthroplasty. Reg Anesth Pain Med. 2005 Sep-Oct;30(5):452-7. doi: 10.1016/j.rapm.2005.05.008. PMID 16135349
- [Background] Kandasami M, Kinninmonth AW, Sarungi M, Baines J, Scott NB. Femoral nerve block for total knee replacement - a word of caution. Knee. 2009 Mar;16(2):98-100. doi: 10.1016/j.knee.2008.10.007. Epub 2008 Nov 28. PMID 19046884
- [Background] Horn JL, Pitsch T, Salinas F, Benninger B. Anatomic basis to the ultrasound-guided approach for saphenous nerve blockade. Reg Anesth Pain Med. 2009 Sep-Oct;34(5):486-9. doi: 10.1097/AAP.0b013e3181ae11af. PMID 19920424
- [Background] Akkaya T, Ersan O, Ozkan D, Sahiner Y, Akin M, Gumus H, Ates Y. Saphenous nerve block is an effective regional technique for post-menisectomy pain. Knee Surg Sports Traumatol Arthrosc. 2008 Sep;16(9):855-8. doi: 10.1007/s00167-008-0572-4. Epub 2008 Jun 24. PMID 18574578
- [Background] Manickam B, Perlas A, Duggan E, Brull R, Chan VW, Ramlogan R. Feasibility and efficacy of ultrasound-guided block of the saphenous nerve in the adductor canal. Reg Anesth Pain Med. 2009 Nov-Dec;34(6):578-80. doi: 10.1097/aap.0b013e3181bfbf84. PMID 19916251

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from the period of 4/16/12-9/4/13 at the Hospital for Special Surgery. Patients were identified on the day of surgery and randomized prior to the start of surgery.
Pre-assignment Details: Patients were excluded prior to randomization if they had contraindications to spinal or epidural anesthesia, had chronic opioid use, pre-existing neuropathies in the limbs, allergies to pre-operative medications, contraindication to assigned nerve blocks, allergy to local anesthetic, American Society of Anesthesia 4-5, and non-English speaking.
Period: Overall Study
Arm/Group | Study Technique Right Leg, Control Technique Left Leg | Study Technique Left Leg, Control Technique Right Leg
Started | 30 | 30
Completed | 29 | 30
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 60
Age, Customized [Mean (Standard Deviation); unit: years] — Age
  years
    Age | 64.41 (7.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale Pain Score
Description: The primary outcome is the postoperative pain in each leg within the first 24 hours postoperatively. VAS pain scores could range from 0 to 10. Higher values represent a worse outcome.
Time Frame: Up to postoperative day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Study Technique: Saphenous Nerve Block: Study Technique: One leg will receive the saphenous nerve block, at the level of the adductor canal. The block will be under ultrasound guidance. The local anesthetic will be 15 ml of 0.5% bupivacaine. All study patients, regardless of study arm will receive combined spinal epidural, with 3 ml of 0.5% bupivacaine as the spinal agent. Epidural local anesthetic, if needed, will consist of 2% lidocaine.
- Control Technique: Femoral Nerve Block: Control Technique: The other leg will receive the femoral nerve block. The block will be under ultrasound guidance. The local anesthetic will be 30 ml of 0.25% bupivacaine. All study patients, regardless of study arm will receive combined spinal epidural, with 3 ml of 0.5% bupivacaine as the spinal agent. Epidural local anesthetic, if needed, will consist of 2% lidocaine.
Arm/Group | Study Technique: Saphenous Nerve Block | Control Technique: Femoral Nerve Block
Number analyzed (Participants) | 59 | 59
units on a scale | 2.81 (2.42) | 2.47 (2.38)

2. Secondary Outcome: Tracking Total Opioid Usage
Time Frame: Up to postoperative day 2
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | All Patients
Number analyzed (Participants) | 59
milligrams | 133.11 (114.53)

3. Secondary Outcome: Preoperative and Postoperative Thigh Muscle Strength in Both Legs
Description: This was measured with a dynamometer to gauge strength.
Time Frame: Up to postoperative day 2
Measure: Mean (Standard Deviation); unit: kilogram-force unit
Arm/Group | Study Technique: Saphenous Nerve Block | Control Technique: Femoral Nerve Block
Number analyzed (Participants) | 59 | 59
kilogram-force unit
  Baseline | 17.06 (10.65) | 17.24 (14.37)
  6-8 h postoperative | 2.86 (3.55) | 2.45 (3.31)
  24 h postoperative | 5.00 (3.68) | 5.08 (4.06)
  48 postoperative | 3.35 (2.62) | 3.76 (3.35)

4. Secondary Outcome: Patient Satisfaction With Nerve Blocks
Description: Rated on a 0-10 scale, with a higher score representing greater satisfaction.
Time Frame: Up to postoperative day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Technique: Saphenous Nerve Block | Control Technique: Femoral Nerve Block
Number analyzed (Participants) | 59 | 59
units on a scale | 8 (2.4) | 8.4 (2.3)

5. Secondary Outcome: Duration of Motor and Sensory Blockade
Time Frame: Up to postoperative day 2
Population: The duration of motor and sensory blockade was not calculated and analyzed, because accurate data regarding block resolution time could not be acquired from patients.
Arm/Group | All Patients
Number analyzed (Participants) | 0

6. Secondary Outcome: Rating the Success of the Nerve Blocks
Time Frame: Up to postoperative day 2
Population: The success of nerve blocks was not collected or analyzed. Instead, muscle strength was collected (data are presented in another table).
Arm/Group | All Patients
Number analyzed (Participants) | 0

7. Secondary Outcome: Postoperative Complications
Time Frame: Up to postoperative day 2
Population: Analysis of postoperative complications was not performed because sufficient data could not be collected regarding the secondary outcome
Arm/Group | All Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The study was monitored for adverse events over the course of 1 year.
Arm/Group | Study Technique: Saphenous Nerve Block | Control Technique: Femoral Nerve Block
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 1/60 | 0/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Technique: Saphenous Nerve Block (N=60) | Control Technique: Femoral Nerve Block (N=60)
Epidural failure (General disorders) | 1 (1) | 0 (0) — Epidural pump for patient malfunctioned

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes